CLINICAL TRIAL: NCT04355195
Title: Quality Contract Prevention of Postoperative Delirium in the Care of Older Patients (QV-POD-2)
Brief Title: Quality Contract: Prevention of Postoperative Delirium in the Care of Older Patients (QV-POD-2)
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: BARMER (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK/CBF), Charite University, Berlin, Germany
Other Study IDs: QV-POD-2
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Delirium in Old Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort before training: 500 patients should be asked to participate in the project in the phase of zero value measurement. The documentation of the routine data before the training phase relates to patients aged ≥70 years, male and female, who are undergoing surgery.
- Cohort after training 1: From October 1st, 2020, the documentation of the routine data will begin after the training phase: 2,500 patients in 12 months, each aged ≥70 years, male and female, who will have surgery until the end of the contract on June 30th, 2023.
- Cohort after documentation of routine data until June 2023: From July 1st, 2023, the documentation of the routine data will go on: 1,700 patients in 12 months, each aged ≥70 years, male and female, who will have surgery until the end of the contract on June 30th, 2028.

SUMMARY:
The project "QV-POD-2" is a prolongation based on "QV-POD-1", which was a quality contract program of the IQTIG - Institute for Quality and Transparency in Health Care. The aim is to improve inpatient care for older patients who are undergoing inpatient surgery and thus to specifically reduce the postoperative risk of delirium. This is achieved through the implementation of evidence-based and consensus-based measures to prevent postoperative delirium in a comprehensive structured concept in routine care. The transparent documentation in an electronic patient file enables the relationships between the symptoms to be depicted in accordance with the clinical circumstances and the genesis of the postoperative delirium to be recorded and treated at an early stage. The content of the additional elements from the routine data (see primary and secondary outcome measures) in QV-POD-2 is analysed internally.

Subproject Retro-Pressure started in August 2022:

Retrospective, exploratory cohort study using electronic anesthesia and hospital records from Jan 1, 2016 to Jan 1, 2020, including patients ≥70 years undergoing surgery with anesthesia. The objective is to quantify associations between intraoperative blood pressure dynamics-variability, rate of change, relative hypo-/hypertension versus baseline, and time-integrated BP (area under/above reference)-and postoperative organ dysfunction Primary endpoints: Emergence delirium incidence (PACU/ITS) based on Nu-DESC scores and CAM-ICU scores; incidence of postoperative acute renal failure (creatinine and urea levels, as well as urine output); intraoperative blood pressure variation*; intraoperative blood pressure variation rate*; intraoperative blood pressure integral* Secondary endpoints: Blood count (hemoglobin and hematocrit values); intraoperative transfusions of blood reserves Addendum from the ethics amendment vote of 25/07/2022

Subproject Delta-Scan started in August 2022:

Evaluation of brain function using "Delta Scan" Primary objective: Evaluation of the prognostic significance of Delta Scan measurements in relation to postoperative delirium Secondary objectives: Examination of the delirium-related predictive relevance of individual influencing factors (directly but also indirectly through Delta Scan values) and examination of the effect of Delta Scan measurements on standard delirium screening methods. Study and control group's Inclusion criteria: Age >= 70 years and major surgery with anesthesia; additional exclusion criterion in the control group: Inclusion in the QV-POD-1 project (receipt of postoperative preventive measures) Addendum from the ethics amendment vote of 25/07/2022

DETAILED DESCRIPTION:
The quality contract of the Charité Universitätsmedizin Berlin QV-POD was contractually extended so that the patients of the Charité Universitätsmedizin Berlin can be offered the preventive measures for delirium for another 5 years (07/01/2023 - 06/30/2028). The continuation of the contract is referred to with the short title QV-POD-2. In terms of content, all preventive measures known from QV-POD will be continued.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 70 years
* male and female patients
* Patients who are insured with BARMER, HEK, KKH, DAK, TK or hkk Health insurances
* Patients eligible for inclusion: by the patient, preoperatively
* Incapacitated patients for inclusion: Written informed consent by a legal representative
* surgery (elective and not elective)

Exclusion criteria:

* Moribund patients
* Not enough language skills

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged ≥70 years, male and female, who are receiving surgery
Sampling Method: Probability Sample
Enrollment: 18100 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Sustainability of implementation rates | Up to 5 years
  QV-POD-2: Sustainability of implementation rates (=Number of patients who underwent delirium screening at least twice a day within the first three days postoperatively / Divisor = All recruited patients) of at least 80% for screening and documentation in the next five years.
Implementation rates | Up to 3 years
  QV-POD-1: Implementation rates (=Number of patients who underwent delirium screening at least twice a day within the first three days postoperatively / Divisor = All recruited patients) of at least 60% for screening and documentation in the first year, at least 70% in the second year and at least 80% in the third year. Addendum to the primary outcome measures from the ethics amendment vote of 25/07/2022)

SECONDARY OUTCOMES:
Sustainability of implementation rates | Up to 5 years
  QV-POD-2: Sustainability of implementation rates (=Number of patients who underwent delirium screening at least twice a day within the first five days postoperatively / Divisor = All recruited patients) of at least 80% for screening and documentation in the next five years
Implementation rates | Up to 5 years
  QV-POD-1: Implementation rates (=Number of patients who underwent delirium screening at least twice a day within the first five days postoperatively / Divisor = All recruited patients) of at least 60% for screening and documentation in the first year, at least 70% in the second year and at least 80% in the third year. Addendum to the secondary outcome measures from the ethics amendment vote of 25/07/2022)
Care level | Up to one year
  The care level is taken from hospital records preoperatively and postoperatively
Routine laboratory | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Routine laboratory markers
Routine vital parameters | The participants are followed up until the end of hospital stay, an expected average of 7 days
Measurement of cholinesterases | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Cholinesterases (point of care testing (POCT) measurements) are measured in the routine
Intraoperative routine data | Time of surgery
Postoperative routine data on the ICU, in the recovery room and normal ward | The participants are followed up until the end of hospital stay, an expected average of 7 days
Drug administration during inpatient treatment | The participants are followed up until the end of hospital stay, an expected average of 7 days
Routine preventive measures against delirium | The participants are followed up until the end of hospital stay, an expected average of 7 days
Intraoperative documented peculiarities in patients with delirium | Time of surgery
Anticholinergic drug intake | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Scale to identify the severity of anticholinergic drugs (Level 0 = no anticholinergic effect, Level 1 = mild anticholinergic effect, Level 2 = moderate anticholinergic effect, Level 3 = severe anticholinergic effect). The sum of all levels of the different drugs gives the total load. Higher total loads of anticholinergic drugs are associated with higher anticholinergic drug load. Minimum of the scale is 0. Maximum depends on the sum of each drug level. The more drugs with anticholinergic effect are taken the higher is the anticholinergic drug load.
Duration of postoperative delirium | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Duration of postoperative delirium in all postoperative patients in normal ward, intensive care unit and recovery room is measured in days (a defined day before the start of the training measures, a defined day after the completion of the training measures). Addendum to the secondary outcome measures from the ethics amendment vote of 25/07/2022)
Incidence of postoperative delirium | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Incidence of postoperative delirium in all postoperative patients in normal ward, intensive care unit and recovery room after validated delirium screening tool at two points in time (a defined day before the start of the training measures, a defined day after the completion of the training measures).
Electroencephalography (EEG) measurement | During the duration of surgery, an expected average of 2 hours
  Objective non-invasive EEG is measured intraoperatively
Infections | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Infections according to surgical site infections (SSI) and according to the US Centers for Disease Control and Preventions (CDC).
Quality of life 1 | Up to three months
  Health related quality of life is measured by EQ-5D-5L
Post Intensive Care Syndrome (PICS) | Up to one year
  The composite outcome measure "PICS" of the patient is measured according to Needham et al 2012: new impairment or worsening of health after intensive care unit stay and at the same time clinically significant distress in at least one of the following outcome measurement instruments: Patient Health Questionnaires (PHQ-9, PHQ-8, PHQ-4), Generalized Anxiety Disorder Scales (GAD-2 and GAD-7), Impact of Event Scale Revised (IES-R), MiniCog, Animal Naming Test, Trail Making Test (TMT-A, TMT-B), Repeatable Battery for the Assessment of Neuropsychological Satus (RBANS), Timed Up-and-Go (TUG), Handgrip Strength, EQ-5D-5L, subjective assessment NRS, WHO Disability Assessment Schedule (WHODAS), Short Physical Performance Battery (SPPB). The Measurement will be performed, when patients present to the outpatient clinic for follow-up examinations. Optionally, the measurement can also be performed via outpatient structures or during a home visit.
Postoperative complications | The participants are followed up until the end of hospital stay, an expected average of 7 days
  To evaluate the presence or development of postoperative organ complications during inpatient care
Analgesia consumption | Up to one year
  Concomitant pain medication is recorded
Postoperative cognitive impairment | Up to three months
  Telephone or Video or questionnaire Follow up is offered to every patient with POD three months and one year after their surgery intervention. The aim of Telephone or Video or questionnaire Follow up is to assess to present Neurocognitive disorder (NCD).The Follow up screening tool is based on DSM 5 diagnostic criteria for "mild cognitive disorder". If one of the diagnostic criteria applies, we recommend to visit a neuropsychologist/ memory clinic recommend to visit a neuropsychologist/ memory clinic.
Depression | Up to one year
  Depression is measured by Patient Health Questionnaire-8 (PHQ-8).This scale encompasses eight questions, which can be answered with not at all (0), several days (1), more than half the days (2) and nearly every day (3). The score is the sum of the 8 items. The minimum score is 0 (best outcome) and the heights 24 (worse outcome).
Anxiety | Up to one year
  Anxiety is measured by Generalized Anxiety Disorder Scale-7 (GAD-7).The Assessment method has seven items; each can be answered with not at all (0), several days (1), more than half the days (2) and nearly every day (3). The score is the sum of all items. The minimum and maximum score are 0 (better outcome) and 21 (worse outcome) respectively.
Physical function | Up to one year
  Physical health is measured by the sum scores of the following outcome measurement instruments: Timed Up-and-Go (TUG), Handgrip Strength, 2-Minute Walk Test (2-MWT), Short Physical Performance Battery (SPPB).
Intensive care unit length of stay | Participants will be followed for the duration of intensive care stay, an expected average of 2 days
  Intensive care unit length of stay is measured in days
Hospital length of stay | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Hospital length of stay is measured in days
Pain levels | Up to one year
  Pain levels are measured with validated subjective/objective pain scores.
Disability 1 | Up to one year
  Disability 1 is measured by Instrumental activities of daily living scale.This scale has 8 categories (ability to use telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility for own medications, ability to handle finances). Each has different levels of functioning with a score assigned. The patient circles the item that most closely describes its functional level. The lowest score is 0 (better outcome) and the highest is 8 (worse outcome).
Disability 2 | Up to one year
  Disability 2 is measured by Timed up and go test.
Disability 3 | Up to one year
  Disability 3 is measured by hand grip strength test
Anxiety-Score | Up to one year
  Faces Anxiety Scale score
Sedation | Up to one year
  Sedation is measured with the Richmond Agitation and Sedation Scale (RASS)
Person's level of consciousness | The participants are followed up until the end of hospital stay, an expected average of 7 days
  The Glasgow Coma Scale (GCS) is a clinical scale used to reliably measure a person's level of consciousness after a brain injury. The GCS assesses a person based on their ability to perform eye movements, speak, and move their body. These three behaviors make up the three elements of the scale: eye, verbal, and motor. A person's GCS score can range from 3 (completely unresponsive) to 15 (responsive). This score is used to guide immediate medical care after a brain injury (such as a car accident) and also to monitor hospitalized patients and track their level of consciousness.
  Lower GCS scores are correlated with higher risk of death.
Permanent medication | Up to one year
  Medication at three months compared to baseline is assessed.
Frailty status | Up to one year
  Frequency of frailty is measured by modified Fried criteria (category 1 +2 = pre-frail, category 3 -5 = frail)
Postoperative oral ingestion | The participants are followed up until the end of hospital stay, an expected average of 7 days
  Ingestion is measured by the amount of fluids and solid food.
Barthelindex | Up to one year
  Score of the Barthel Index ranging from 0 to 100 were collected when 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
  Score was reported as mean score of the Barthel Index.
Patient-related outcome measures (PROMS) | Up to one year
  Different tools and questionnaires are combined to measure Patient-related outcome.
Patient-related experience measures (PREMS) | Up to one year
  Patient-reported experiences of health care are measured with a questionnaire.
Therapy recommendations | Up to one year
  Therapy recommendations are documented from patient records.
Survival | Up to one year
  Survival is measured in Patients form QV-POD-2 within 1 year; Survival is measured in patients from QV-POD-1 until 3 months (addendum to the secondary outcome measures from the ethics amendment vote of 28/08/2025).

OTHER OUTCOMES:
Preoperative routine data | At baseline
  Preoperative routine data are medical history, diagnoses, medication, etc.
Patient-specific characteristics | At baseline
  Patient-specific characteristics of patients with delirium
Preoperative risk score for delirium | At baseline
  Development of a risk model with different influencing factors of delirium
Preoperative sober times | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Department of Anesthesiology and Intensive Care Medicine (CBF), Charité - Universitätsmedizin Berlin, Berlin
  - Department of Anesthesiology and Intensive Care Medicine (CCM/CVK) Berlin, Carité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yurek F, Zimmermann JD, Weidner E, Hauss A, Dahnert E, Hadzidiakos D, Kruppa J, Kiselev J, Sichinava N, Retana Romero OA, Hoff L, Morgeli R, Junge L, Scholtz K, Piper SK, Gruner L, Harborth AEM, Eymold L, Gulmez T, Falk E, Balzer F, Treskatsch S, Hoft M, Schmidt D, Landgraf F, Marschall U, Holscher A, Rafii M, Spies C. Quality contract 'prevention of postoperative delirium in the care of elderly patients' study protocol: a non-randomised, pre-post, monocentric, prospective trial. BMJ Open. 2023 Mar 6;13(3):e066709. doi: 10.1136/bmjopen-2022-066709. PMID 36878649